CLINICAL TRIAL: NCT00865878
Title: A Randomized, Evaluator-Blinded, Parallel Group Comparison of PDT With Levulan Topical Solution + Blue Light vs Levulan Topical Solution Vehicle + Blue Light for the Treatment of AK and Reduction of New NMSC in Organ Transplant Recipients
Brief Title: ALA-PDT Versus Vehicle PDT for Treatment of AK and Reduction of New NMSC in Solid Organ Transplant Recipients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Orphan Drug Designation for this indication not granted
Sponsor: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DUSA-CP0104
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Actinic Keratoses; Skin Neoplasms
Keywords: Actinic Keratoses; Skin Neoplasms; Photodynamic Therapy; Transplants
MeSH Terms: conditions — Keratosis, Actinic; Skin Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Topical Levulan Kerastick containing 20% aminolevulinic acid HCL (ALA) will be applied to the entire scalp OR both forearms 90 +/- 30 minutes prior to blue light treatment for 16 minutes and 40 seconds.
  Interventions: Drug: Aminolevulinic Acid
- 2 (Placebo Comparator): Kerastick containing vehicle ingredients only (VEH) will be applied to the entire scalp OR both forearms 90 +/- 30 minutes prior to blue light treatment for 16 minutes 40 seconds.
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: Aminolevulinic Acid — 20% aminolevulinic acid HCL (ALA) applied topically for 90 +/- 30 minutes prior to treatment with 10 j/cm2 blue light. Up to nine (9) ALA-PDT treatments will be given: The initial four (4) treatments will be given at 4-5 week intervals, with the remaining five (5) treatments given every 6 +/-1 weeks.
  Other Names: Levulan
  Arms: 1
Other: Vehicle — Vehicle ingredients only (VEH) applied topically for 90 +/- 30 minutes prior to treatment with 10 j/cm2 blue light. Up to nine (9) VEH-PDT treatments will be given: The initial four (4) treatments will be given at 4-5 week intervals, with the remaining five (5) treatments given every 6 +/-1 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to determine and compare the safety and efficacy of broad area photodynamic therapy with aminolevulinic acid (ALA-PDT) versus vehicle PDT (VEH-PDT) in the treatment of actinic keratoses (AK) and reduction of new non-melanoma skin cancer (NMSC) of the scalp or both forearms in solid organ transplant recipient subjects receiving chronic immunosuppressive therapy.

DETAILED DESCRIPTION:
This is a Phase II multicenter, randomized, evaluator-blinded, vehicle-controlled, parallel group study of photodynamic therapy in organ transplant recipient subjects for treatment of AK and the reduction of new NMSC.

Subjects will be randomized to one of the following two treatment groups (1:1) to receive topical Levulan® Kerastick® containing 20% aminolevulinic acid HCL (ALA, active study drug) or the Kerastick® containing vehicle ingredients only (VEH).

* Group 1 will have ALA applied to the entire scalp OR both forearms 90 +/- 30 minutes prior to BLUE light treatment for 16 minutes 40 seconds
* Group 2 will have VEH applied to the entire scalp OR both forearms 90 +/- 30 minutes prior to BLUE light treatment for 16 minutes 40 seconds

Treatment Area (scalp or both forearms) must have had at least 2 NMSC in the past 12 months, and must include a continuous 25 cm2 Target Area containing a minimum of 3 AKs, to be eligible for treatment

Each subject may receive up to nine treatments. The initial four (4) ALA-PDT/VEH-PDT treatments will be given at 4-5 week intervals, with the remaining five (5) treatments given every 6 +/-1 weeks. Post-treatment follow-up visit will be scheduled to occur 4 weeks after the subject's final PDT.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or non-pregnant female organ transplant (kidney, liver, pancreas, lungs, heart or combinations thereof) recipient outpatient 18 years of age or older. Females must be post-menopausal, surgically sterile or using a medically acceptable form of birth control, with a negative urine pregnancy test at the Baseline visit.
2. Subject has provided written and verbal informed consent.
3. Subject has at least 3 actinic keratosis lesions in a continuous 25 cm2 Target Area within the selected anatomic treatment site (scalp or forearm).
4. Subject has a history of a minimum of 2 NMSC on the treatment area of interest (scalp OR both forearms) in the past 12 months
5. Subject is currently receiving standard active pharmacologic immunosuppression
6. Subject is willing to comply with study instructions and return to the clinic for required visits.
7. Subject has Fitzpatrick skin type I-IV.

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject has a history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis.
3. Subject has any skin pathology or condition, in the investigator's opinion, that could interfere with the evaluation of the test product or requires the use of interfering topical or systemic therapy.
4. Subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
5. Subject is currently enrolled in an investigational drug (including experimental immunosuppressive agents containing new chemical entities) or device study. Novel combinations of and alternative dosing regimens of approved immunosuppressive agents are allowed.
6. Subject has received an investigational drug (including experimental immunosuppressive agents containing new chemical entities) or been treated with an investigational device within 30 days prior to the initiation of treatment (baseline). Novel combinations of and alternative dosing regimens of approved immunosuppressive agents are allowed.
7. Subject is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
8. Subject may be unreliable for the study including subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits.
9. Subject has a known sensitivity to one or more of the vehicle components (ethyl alcohol, isopropyl alcohol, laureth 4, polyethylene glycol).
10. Subject has active recurrent herpes simplex labialis infection in the treatment area with an outbreak within the last 12 months and will not be placed on antiviral prophylaxis as specified in the protocol.
11. Subject has used any of the following topical preparations on the selected Treatment Area (scalp OR both forearms):

    * Keratolytics including urea (greater than 5%), alpha hydroxyacids [e.g. glycolic acid, lactic acid, etc. greater than 5%], salicylic acid (greater than 2%) within 2 days of initiation of treatment.
    * 5-FU, cryotherapy, diclofenac, imiquimod or other treatments for AK within 2 weeks of initiation of treatment
    * Retinoids, including tazarotene, adapalene, tretinoin, retinol, within 4 weeks of the initiation of treatment.
    * Microdermabrasion, laser ablative treatments, ALA-PDT or chemical peels within 8 weeks of the initiation of treatment.
    * Two or more ALA PDT treatments in the past 6 months
12. Subject has used systemic retinoid therapy within 6 months of the initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of Skin Cancers within the Treatment Area | entire study
AK Lesions Counts/Surface Area | Visits 1,3,5,7,9,11,13,15,17,19
Investigator Global Assessment | Visits 1,3,5,7,9,11,13,15,17,19

SECONDARY OUTCOMES:
Subject Acceptability of Treatment | End of Study
Tolerability Parameters | Each Visit

CONTACTS AND LOCATIONS:
Overall Officials: Stuart L Marcus, MD, PhD, Study Director — Sponsor GmbH
Locations (7):
- United States (7):
  - University of California, Irvine, Irvine, California
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - The Mount Sinai Medical Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee